CLINICAL TRIAL: NCT02810821
Title: Association Between Serum Gonadal Hormone, Gonadotropin and Cardiovascular Events
Brief Title: Gonadal Hormone, Gonadotropin and Cardiovascular Events
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jia-jun Zhao, Professor, Shandong Provincial Hospital
Other Study IDs: 20140722
Record Dates: First submitted 2016-06-11; First posted 2016-06-23 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Aging; Menopause
Keywords: Gonadal hormones; Gonadotropins; Cardiovascular diseases; Lipids; Obesity; Atherosclerosis; Glucose metabolism disorders; Metabolic syndrome; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Atherosclerosis; Glucose Metabolism Disorders; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum，Plasma and Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- female, premenopause: Women with regular menstrual cycles in normal range (22-35 days) for the previous three cycles.
- female, perimenopause: Peri-menopause was defined as the presence of menses within the past 3 months with a decrease in cycle predictability in the year preceding examination or 3-11 months of amenorrhea. To investigate the association between serum FSH and cholesterol levels independent of E2, we further selected peri-menopausal subjects with the presence of menses within the past 3 months with a decrease in cycle predictability in the year preceding examination because their E2 levels have been reported to be similar to those in pre-menopause.
- Serum FSH level Quartile 1: Serum FSH level: <6.95 mIU/mL
- Serum FSH level Quartile 2: Serum FSH level: 6.95-10.87 mIU/mL
- Serum FSH level Quartile 3: Serum FSH level: 10.88-25.45 mIU/mL
- Serum FSH level Quartile 4: Serum FSH level: >25.45 mIU/mL

SUMMARY:
Deficiency in gonadal hormone has been considered to play a role in ageing related increased incidence of cardiovascular events. But the mechanism has not been fully elucidated. On the other hand, the dramatic increase in gonadotropin level didn't drew much attention when talking about the increased risk of cardiovascular disease during menopausal transition. This study aim to investigate the association between gonadal hormone, gonadotropin and long-term cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with intact uterus and at least one ovary
* Aged of 18 to 75 years old;

Exclusion Criteria:

* Pregnancy or lactation women;
* Presence of pituitary/hypothalamic disorders, polycystic ovarian syndrome or other endocrinal and metabolic disorders that known to compromise hypothalamic-pituitary-gonadal function;
* Receiving psychotropic or hormonal medications including hormonal contraception and hormone therapies;
* Taking lipid-lowering agents or hypoglycemic agents and other drugs that known to influence cardiovascular health;
* Obviously poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged of 18 to 75 years old. Part of the subjects (aged 40 years or more) were selected from REACTION study that was conducted from April,1, 2011 through May 30, 2012, aiming to investigate the epidemiology of metabolic diseases across China. The younger participants were recruited since July 1, 2014.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2011-07; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Rate of first cardiovascular disorder events | Measured after 10 years of follow-up
  Total incidence rate from cardiovascular disorder over a given period of time
Cardiovascular disease mortality | Measured after 10 years of follow-up
  Total deaths from cardiovascular disease over a given period of time
All-cause mortality | Measured after 10 years of follow-up
  Total deaths from all causes over a given period of time

SECONDARY OUTCOMES:
Change in serum lipid levels | Measured at baseline, and every 2 years during the 10-year follow-up period
  Include triglycerides、cholesterol、 low density lipoprotein cholesterol、 high density lipoprotein cholesterol.
Change in thickness of blood vessel wall | Measured at baseline, and every 2 years during the 10-year follow-up period
  The mean carotid Intima media thickness showed the early risk of atherosclerotic cardiovascular diseasean. the subclinical atherosclerosis was defined as the mean carotid Intima media thickness ≥0.78mm.
Number of participants that diagnosed with metabolic syndrome | Measured at baseline, and every 2 years during the 10-year follow-up period
  Metabolic syndrome refers to the pathological state in which protein, fat, carbohydrate and other substances in human body have metabolic disorders. It is a group of complex metabolic disorders and a risk factor leading to cardiovascular and cerebrovascular diseases of diabetes.
Number of participants that diagnosed with non-alcoholic fatty liver disease | Measured at baseline, and every 2 years during the 10-year follow-up period
  A clinicopathological syndrome characterized by excessive deposition of fat in liver cells due to alcohol and other clearly damaging factors is excluded

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhao, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

REFERENCES:
- [Background] Guo Y, Zhao M, Bo T, Ma S, Yuan Z, Chen W, He Z, Hou X, Liu J, Zhang Z, Zhu Q, Wang Q, Lin X, Yang Z, Cui M, Liu L, Li Y, Yu C, Qi X, Wang Q, Zhang H, Guan Q, Zhao L, Xuan S, Yan H, Lin Y, Wang L, Li Q, Song Y, Gao L, Zhao J. Blocking FSH inhibits hepatic cholesterol biosynthesis and reduces serum cholesterol. Cell Res. 2019 Feb;29(2):151-166. doi: 10.1038/s41422-018-0123-6. Epub 2018 Dec 17. PMID 30559440
- See also: NCBI link — https://pubmed.ncbi.nlm.nih.gov/30559440/